CLINICAL TRIAL: NCT06585163
Title: A Phase 1, Randomized, Double-blind, Crossover Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of QEV-817 Oral Suspension in Healthy Volunteers
Brief Title: Study to Investigate the Safety, Tolerability and Pharmacokinetics of QEV-817 Oral Suspension
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Quivive Pharma, Inc. (Industry)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Supportive Care
Other Study IDs: QEV-817-101; 5R44DA055336 (NIH)
Record Dates: First submitted 2024-09-01; First posted 2024-09-05 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-09

CONDITIONS: Healthy
MeSH Terms: interventions — Hydrocodone; Doxapram

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized to receive A) hydrocodone and B) hydrocodone + doxapram in one of two possible sequences (ie. A followed by B or B followed by A).
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sequence A - Hydrocodone alone followed by combined (hydrocodone + doxapram) (Experimental): Subjects randomized to Sequence A will first receive a single oral administration of hydrocodone bitartrate alone on Study Day-2 and then receive a combination of hydrocodone bitartrate and doxapram hydrocholoride on study Day-4 (after a 48 hour wash-out).
  Interventions: Drug: Hydrocodone Bitartrate; Drug: Doxapram Hydrochloride
- Sequence B - Combined (hydrocodone + doxapram) followed by hydrocodone alone (Experimental): Subjects randomized to Sequence B will first receive a single combined administration of hydrocodone bitartrate and doxapram hydrocholoride on Study Day-2 and then receive hydrocodone alone on study Day-4 (after a 48 hour wash-out).
  Interventions: Drug: Hydrocodone Bitartrate; Drug: Doxapram Hydrochloride

INTERVENTIONS:
Drug: Hydrocodone Bitartrate — Hydrocodone bitartrate oral suspension
  Other Names: NDC 51634-0014
Drug: Doxapram Hydrochloride — Doxapram hydrocholoride oral suspension
  Other Names: NDC 10920-601

SUMMARY:
This study has been designed to assess the safety, tolerability, and pharmacokinetics of a therapeutic dose of hydrocodone bitartrate with and without an oral dose of doxapram hydrochloride in healthy volunteers who are naltrexone-blocked.

DETAILED DESCRIPTION:
This is a Phase 1, single-center, double-blind, randomized crossover study that will be conducted in male and female healthy volunteers. The study will be conducted at a single site in the US. The study consists of a 28-day Screening Period, a four-day treatment period, and a one-day safety follow-up period.

The study will be conducted in eight (8) healthy male and female subjects. Up to an additional five (5) subjects may be enrolled as alternates to replace dropouts. Subjects will be randomized (1:1) to one of two crossover treatment sequences.

The subjects, Investigators, and site personnel (except site personnel responsible for study treatment preparation) will be blinded to treatment assignments. Subjects will receive either a fixed therapeutic dose of oral hydrocodone alone or in combination with a fixed dose of oral doxapram. Prior to treatment, all subjects will receive naltrexone (opioid antagonist) to block opioid effects (i.e., naltrexone block).

Safety will be evaluated by monitoring the nature, severity, and incidence of adverse events (AEs); and changes from baseline in physical examination, vital signs, 12-lead electrocardiogram (ECG) assessment, pulse oximetry, and clinical laboratory tests.

Pharmacokinetics of both drugs and their primary metabolites will be assessed in plasma samples collected through 24 hours post-dose from all subjects. All enrolled subjects will also be genotyped for CYP2D6 polymorphism status.

ELIGIBILITY:
Key Inclusion Criteria - include but are not limited to:

* Male or female aged 18-55 years, inclusive, on the day of screening.
* Willing to abstain from alcohol and strenuous physical activity (i.e., strenuous, or unaccustomed weightlifting, running, bicycling, etc.) from 48 hours prior to study treatment administration until discharge from the clinical unit and prior to each outpatient visit.
* Have normal laboratory values, as defined per protocol, at screening.
* Absence of cardiac arrythmias, as well as corrected QT interval (QTc) < 450 ms in males and QTc < 460 ms in females based on 12-lead ECG findings at screening.
* Body weight ≥50 kg and body mass index (BMI) within the range of 19-32 kg/m2 (inclusive).
* Has never used opioids for non-therapeutic purposes (i.e., for recreational effects). Subjects with a history of valid medical use under prescription must have not used an opioid for at least three (3) months prior to Day 1.
* Women of childbearing potential (WOCBP), as defined in Section 10.4, must have a negative serum pregnancy test within one (1) week AND a negative urine pregnancy test on Day 2, prior to the start of study treatment; Must not be breastfeeding, lactating, or planning a pregnancy during the study and for at least 32 days (5 half-lives plus 30-days) after the last dose of study intervention
* Postmenopausal females must have a documented serum follicle-stimulating hormone (FSH) level >40 mIU/mL (milli international units per milliliter) at screening to confirm menopause.
* Male participants with female sexual partners who are WOCBP must agree to remain abstinent (complete avoidance of heterosexual intercourse) or use adequate contraceptive methods, defined as use of a condom by the male partner combined with use of a highly effective method of contraception by the female partner, during the treatment period and for at least 92 days (5 half-lives + 90-day spermatogenesis cycle) after the last dose of study intervention; must not donate sperm for at least 92 days (5 half-lives + 90-day spermatogenesis cycle) after the last dose of study intervention.

Exclusion Criteria - include but are not limited to:

* Female subject who is pregnant or lactating.
* Have any vital sign abnormalities as described in the protocol.
* Recreational opioid user who has used opioids for non-therapeutic purposes (i.e., for psychoactive effects) or who is physically dependent on any illicit or prescription opioid, and/or currently participating in a treatment program for individuals with opioid dependence.
* Known allergy or history of significant adverse reaction to hydrocodone or its metabolites, other opioids, or related compounds, doxapram hydrochloride, naltrexone, naloxone, or to any of the excipients in QEV-817.
* History of or currently has hypoventilation syndrome or sleep apnea and is on non-invasive ventilation (e.g., CPAP).
* Clinically meaningful infection/injury/illness within one month prior to screening.
* Active malignancy (excluding squamous or basal cell carcinoma of the skin) within 5 years of screening.
* Subjects with hepatic impairment as defined by screening alanine transaminase (ALT), aspartate transaminase (AST) or total bilirubin >3× upper limit of normal (ULN).
* Subjects with renal impairment as defined by screening estimated creatinine clearance/eGFR (estimated glomerular filtration rate) using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation is <60 mL/min/1.73 m2.
* Donation of blood (>450 mL) or significant blood loss within 56 days.
* Current (or recent history of) psychiatric illness or mental impairment.
* Clinically meaningful current (or history of) unstable chronic disease; medical abnormality; or significant cardiovascular (including significant cardiovascular impairment, uncompensated heart failure, severe coronary artery disease, severe hypertension), endocrine, gastrointestinal, neurological disorder (including cognitive disorders); or metabolic disease.
* Currently active (or history of) epilepsy, seizure disorder, serious head injury, cerebral vascular accident, or cerebral edema.
* Current treatment with monoamine oxidase inhibitors (MAOIs), tricyclic antidepressants, sympathomimetic drugs, neuromuscular blocking agents, narcotics, antihistamines, antipsychotics, antianxiety agents, or other central nervous system (CNS) depressants.
* Use of any prescription or over the counter (OTC) medications including food supplements and herbal medications (e.g., St. John's wort), with the exception of contraceptive medications or a daily multivitamin, within fourteen (14) days prior to study treatment administration. Use of CYP3A4 inhibitors or inducers is prohibited within 28 days prior to the first treatment and throughout the treatment and follow-up periods.
* A positive urine drug, cotinine, or alcohol test at screening, excluding tetrahydro-cannabinol (THC) or cannabinoid metabolites.
* Smokers or use of tobacco-containing products within 6 weeks of study drug administration.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Treatment-Emergent Adverse Events (TEAEs) | Day 1 to Day 5
  Incidence, nature, and severity of TEAEs
Number of Participants with Abnormal Laboratory Assessments, 12-Lead Electrocardiogram (ECG), and Vital Signs | Day 1 to Day 5
  Changes from baseline in physical examination, vital signs, 12-lead ECG assessment and pulse oximetry

SECONDARY OUTCOMES:
Plasma PK Parameters (Cmax) | Day 2 and Day 4
  Maximal plasma concentrations for hydrocodone and doxapram
Plasma PK Parameters (AUC0-inf) | Day 2 and Day 4
  Plasma area under the curve for hydrocodone and doxapram
Plasma PK Parameters (Tmax) | Day 2 and Day 4
  Time to maximal plasma concentrations for hydrocodone and doxapram

CONTACTS AND LOCATIONS:
Overall Officials: Ryu Komatsu, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Main Campus, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results to be reported, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: Anyone who wishes to access the data for any purpose.